CLINICAL TRIAL: NCT01840540
Title: Phase I Study of Autologous Mesenchymal Stem Cells in the Treatment of Atherosclerotic Renal Artery Stenosis
Brief Title: MSC for Occlusive Disease of the Kidney
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen C. Textor, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-009298
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Atherosclerotic Renal Artery Stenosis; Ischemic Nephropathy; Renovascular Hypertension
Keywords: renal artery stenosis; renovascular hypertension; ischemic nephropathy; chronic kidney disease
MeSH Terms: conditions — Hypertension, Renovascular; Renal Artery Obstruction; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- infusion of autologous mesenchymal stem cells (Experimental): Patients will undergo a subcutaneous fat biopsy for expansion of mesenchymal stromal (stem) cells (MSC) in the Human Cell Therapy Laboratory. Patients will be admitted to the inpatient Clinical Research Unit of the Mayo Clinic Center for 3 days prior to treatment, for pre-infusion tests. Renal angiography will be performed to deliver a single intra-arterial dose of MSC's into one affected kidney. Patients will be observed for 24 hours for acute adverse events. Patients will have remote visits at 1 week, 4 weeks,8 weeks, and 6 months. At 3 months, patients will return for repeat evaluation of kidney function, blood flow and structural alterations within the clinical research unit at St. Mary's Hospital, Rochester, Minnesota. Thereafter, health assessment and blood draws will be repeated at 12 and 24 months with urinary cytology and MRI.
  Interventions: Drug: Arterial infusion of autologous mesenchymal stem cells

INTERVENTIONS:
Drug: Arterial infusion of autologous mesenchymal stem cells
  Other Names: MSC

SUMMARY:
To determine the safety and toxicity of intra-arterial infused autologous adipose derived mesenchymal stromal (stem) cells in patients with vascular occlusive disease of the kidney.

DETAILED DESCRIPTION:
Individuals with unilateral arterial occlusive disease will be treated to injured kidney with autologous cells.

ELIGIBILITY:
4.1 Inclusion Criteria

1. Are between ages 40 and 80 years old.
2. Advanced vascular occlusive disease (atherosclerosis) affecting one or both kidneys: defined as a) loss of parenchymal volume and renal blood flow (measured by MDCT as previously described (17) and/or duplex ultrasound velocity above 300 cm/sec to the affected kidney to be infused with MSC's.
3. Have serum creatinine below 2.5 mg/dL
4. Have no-contraindications to angiography: severe contrast allergy
5. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
6. Ability to comply with protocol
7. Competent and able to provide written informed consent

4.2 Exclusion Criteria

1. Advanced CKD: Stage 5 (two kidney eGFR < 15 ml/min/1.73 m2) contralateral renal artery occlusion/stenosis above 75% or ESRD requiring dialysis
2. Clinically significant abnormalities on laboratory examination, including Bilirubin (> 2 x normal), platelets (<100 thousand), potassium (>5.5 mEq/L), and sodium (<130 mEq/L), ALT or AST more than 2 x normal, Prothrombin time (INR>1.4), Hemoglobin <10.0 g/dL.
3. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure) that would, in the opinion of the investigators, compromise the safety of the patient.
4. Specific exclusions:

   1. Clinical history of deep vein thrombosis within three months of MSC administration
   2. Uncontrolled hypertension (Systolic BP >180 mmHg despite therapy)
   3. Active infection
   4. Reduced ejection fraction (below 30%)
   5. Evidence of hepatitis B,C, or HIV
   6. Diabetes treated with insulin and/or glucose lowering agents
   7. Anemia (Hgb<10 g/dL)
   8. Regular use of potentially renotoxic drugs, e.g. non-steroidal anti-inflammatory agents (NSAID's): (>2 x weekly)
5. History of cancer including melanoma (with the exception of localized skin cancers)
6. Investigational drug exposure within thirty (30) days of baseline
7. Beck's depression score above 16
8. Pregnant or breast feeding.
9. History of clinically significant auto-immunity or any previous example of fat-directed autoimmunity

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Renal blood flow and function in the treated kidneys. | 2 years
  Individual kidney blood flow, measured by multidetector CT contrast transit times, will be measured before and after MSC infusion.

SECONDARY OUTCOMES:
Level of kidney function. | 2 years
  Level of kidney function will be assessed as glomerular filtration rate by iothalamate clearance. Tissue oxygenation within each kidney will be measured by Blood Oxygen Level Dependent (BOLD) magnetic resonance.

OTHER OUTCOMES:
Blood pressure levels. | 2 years
  Blood pressure will be assessed by oscillometric measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Textor, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Camilleri ET, Gustafson MP, Dudakovic A, Riester SM, Garces CG, Paradise CR, Takai H, Karperien M, Cool S, Sampen HJ, Larson AN, Qu W, Smith J, Dietz AB, van Wijnen AJ. Identification and validation of multiple cell surface markers of clinical-grade adipose-derived mesenchymal stromal cells as novel release criteria for good manufacturing practice-compliant production. Stem Cell Res Ther. 2016 Aug 11;7(1):107. doi: 10.1186/s13287-016-0370-8. PMID 27515308